CLINICAL TRIAL: NCT01391962
Title: A Phase II Trial In Which Patients With Metastatic Alveolar Soft Part Sarcoma Are Randomized to Either Sunitinib or Cediranib Monotherapy, With Cross-Over at Disease Progression
Brief Title: Sunitinib or Cediranib for Alveolar Soft Part Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 110200; 11-C-0200
Record Dates: First submitted 2011-07-09; First posted 2011-07-12 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sarcoma, Alveolar Soft Part
Keywords: Pharmacodynamics; VEGF Inhibitor; Alveolar Soft Part Sarcoma; Anti-Angiogenesis; Gene Expression Profiling
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part | interventions — cediranib; Sunitinib; Prochlorperazine; Promethazine; Diphenhydramine; Benzodiazepines; Diazepam; Estazolam; Flurazepam; Lorazepam; Filgrastim; sargramostim; atropine sulfate-diphenoxylate hydrochloride drug combination; Diphenoxylate; Loperamide; Vitamin B 6; Pyridoxine; Petrolatum; Acetaminophen; Thyroxine; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I - Cediranib (30 mg) or Sunitinib Malate (37.5 mg) Orally (Experimental): Patients will be randomized to receive cediranib (30 mg) or sunitinib malate (37.5 mg) orally, once a day in 28-day cycles.
  Interventions: Drug: Cediranib; Drug: Sunitinib; Other: Prochlorperazine; Other: Promethazine; Other: Benzodiazepine; Other: Filgrastim; Other: Sargramostim; Other: Lomotil; Other: Loperamide; Other: Vitamin B6; Other: Aquaphor; Drug: Acetaminophen; Drug: Levothyroxine; Drug: Warfarin
- Part II - Cross Over (Experimental): At the time of disease progression, patients will cross over to the other treatment arm after a 2-week wash-out period.
  Interventions: Drug: Cediranib; Drug: Sunitinib; Other: Prochlorperazine; Other: Promethazine; Other: Benzodiazepine; Other: Filgrastim; Other: Sargramostim; Other: Lomotil; Other: Loperamide; Other: Vitamin B6; Other: Aquaphor; Drug: Acetaminophen; Drug: Levothyroxine; Drug: Warfarin

INTERVENTIONS:
Drug: Cediranib — Cediranib, a small molecule inhibitor of vascular endothelial growth factor (VEGF) receptor tyrosine kinases, is showing preliminary evidence of activity in patients with alveolar soft part sarcoma (ASPS).
  Other Names: AZD2171 maleate; Recentin; AXD2171
Drug: Sunitinib — Sunitinib, a small molecule inhibitor of vascular endothelial growth factor (VEGF) receptor tyrosine kinases, is showing preliminary evidence of activity in patients with alveolar soft part sarcoma (ASPS).
  Other Names: Sutent; SU11248; SU011248
Other: Prochlorperazine — 10mg every 6 hours orally as needed for nausea,
  Other Names: Compro
Other: Promethazine — 12.5-25mg intravenous every 6 hours as needed for nausea.
  Other Names: Phenadoz; Phenergan; Promethegan
Other: Benzodiazepine — If promethazine is inadequate, add benzodiazepine until acute nausea is controlled.
  Other Names: Valium; Diazepam; Estazolam; ProSom; Flurazepam; Dalmane; Lorazepam; Ativan
Other: Filgrastim — Therapeutic use per investigator's discretion according to American Society of Clinical Oncology (ASCO) guidelines.
  Other Names: Neupogen
Other: Sargramostim — Therapeutic use per investigator's discretion according to American Society of Clinical Oncology (ASCO) guidelines.
  Other Names: Leukine
Other: Lomotil — 2.5mg plus atropine sulfate 0.025mg/tablet dosed according to package insert.
  Other Names: Diphenoxylate hydrochloride (HCL)/atropine
Other: Loperamide — 4mg by mouth (PO) after first unformed stool with 2mg PO every 2 hours as long as unformed stools continue.
  Other Names: Imodium; Diamode; Anti-Diarrheal (loperamide)
Other: Vitamin B6 — 50-150mg orally each day for hand-foot syndrome.
  Other Names: Pyridoxine
Other: Aquaphor — Topical emollient for hand-foot syndrome.
Drug: Acetaminophen — Analgesic for hand foot syndrome as needed.
  Other Names: Tylenol; Ofirmev; FeverAll
Drug: Levothyroxine — Replacement therapy for participants with increases in thyroid-stimulating hormone.
  Other Names: Synthroid; Tirosint; Unithroid
Drug: Warfarin — 2mg daily for prophylaxis of thrombosis.
  Other Names: Coumadin

SUMMARY:
Background:

* Alveolar soft part sarcoma (ASPS) is a rare, highly vascular tumor accounting for less than 1% of soft tissue sarcomas. There is no effective systemic treatment for patients with metastatic ASPS. Little is known with regards to relevant molecular markers as potential therapeutic targets.
* Cediranib (AZD2171) and sunitinib (SU011248), oral small molecule inhibitors of vascular endothelial growth factor (VEGF) receptor tyrosine kinases, are showing preliminary evidence of activity in patients with ASPS.

Objectives:

* Part I: Determine the objective response rate (ORR) of single-agent cediranib and single-agent sunitinib malate in patients with advanced ASPS.
* Part II: Determine the ORR of cediranib in patients who progress on the sunitinib arm, and determine the ORR of sunitinib in patients who progress on the cediranib arm.
* Determine the progression-free survival (PFS) at 24 weeks for single-agent cediranib and

single-agent sunitinib malate in patients with advanced ASPS.

Eligibility:

* Patients aged greater than or equal to 16 years with histologically or cytologically confirmed metastatic ASPS.
* Patients must show evidence of objective disease progression per Response evaluation criteria in solid tumors (RECIST)v1 on scans within the 3-month period immediately preceding enrollment. Both scans used to determine disease progression should have been obtained within this 6-month period.
* Patients with newly diagnosed, unresectable, measurable, metastatic ASPS who show clinical evidence of disease progression will be eligible.
* Patients must not have received treatment with any VEGF receptor tyrosine kinase inhibitor (e.g., cediranib, sunitinib, pazopanib, sorafenib); however, prior treatment with bevacizumab is allowed.

Design:

* Part I: Patients will be randomized to receive cediranib (30 mg) or sunitinib malate (37.5 mg) orally, once a day in 28-day cycles.
* Part II: At the time of disease progression, patients will cross over to the other treatment arm after a 2-week wash-out period.
* Appropriate anatomic imaging studies will be performed at baseline and every 2 cycles for restaging.
* The study will be conducted using an optimal two-stage design to rule out an unacceptably low 15% clinical response rate (PR+CR) in favor of a modestly high response rate of 40%.

The study will initially enroll 10 evaluable patients in each arm. If 0 or 1 of the 10 patients has a clinical response, then no further patients will be accrued. If 2 or more the first 10 patients have a response, then accrual continues to a total of 22 patients in each arm.

DETAILED DESCRIPTION:
Background:

* Alveolar soft part sarcoma (ASPS) is a rare, highly vascular tumor accounting for less than 1% of soft tissue sarcomas. There is no effective systemic treatment for patients with metastatic ASPS. Little is known with regards to relevant molecular markers as potential therapeutic targets.
* Cediranib (AZD2171) and sunitinib (SU011248), oral small molecule inhibitors of vascular endothelial growth factor (VEGF) receptor tyrosine kinases, are showing preliminary evidence of activity in patients with ASPS.

Objectives:

* Part I: Determine the objective response rate (ORR) of single-agent cediranib and single-agent sunitinib malate in patients with advanced ASPS.
* Part II: Determine the ORR of cediranib in patients who progress on the sunitinib arm and determine the ORR of sunitinib in patients who progress on the cediranib arm.
* Determine the progression-free survival (PFS) at 24 weeks for single-agent cediranib and single-agent sunitinib malate in patients with advanced ASPS.

Eligibility:

Status Update: Patients enrolled after Amendment G (version dated 08/16/2013), will be evaluated and compared to the first 13 patients by the study statistician and the Principal Investigator. Patients with newly diagnosed ASPS with clinical evidence of disease progression will also be assessed separately.

* Patients aged greater than or equal to 16 years with histologically or cytologically confirmed metastatic ASPS.
* Patients must show evidence of objective disease progression per Response Evaluation Criteria in Solid Tumors (RECIST)v 1 on scans within the 3-month period immediately preceding enrollment. Both scans used to determine disease progression should have been obtained within this 6-month period.
* Patients with newly diagnosed, unresectable, measurable, metastatic ASPS who show clinical evidence of disease progression will be eligible.
* Patients must not have received treatment with any VEGF receptor tyrosine kinase inhibitor (e.g., cediranib, sunitinib, pazopanib, sorafenib); however, prior treatment with bevacizumab is allowed.

Design:

* Two sets of patients will be enrolled and assessed in separate cohorts: a) patients with non-newly diagnosed ASPS and b) patients with newly diagnosed ASPS
* Part I: Patients will be randomized to receive cediranib (30 mg) or sunitinib malate (37.5 mg) orally, once a day in 28-day cycles. As of May 6, 2019, we have closed the cediranib arm of the newly diagnosed ASPS cohort due to inadequate activity per the statistical plan; all newly diagnosed ASPS patients will be assigned to the sunitinib malate treatment arm.
* Part II: At the time of disease progression, patients will cross over to the other treatment arm after a 2-week wash-out period. As of May 6, 2019, patients in the newly diagnosed ASPS cohort are not eligible to cross over to the cediranib treatment arm, which was closed due to inadequate activity.
* Appropriate anatomic imaging studies will be performed at baseline and every 2 cycles for restaging.
* The study will be conducted using an optimal two-stage design to rule out an unacceptably low 15% clinical response rate partial response + complete response (PR+CR) in favor of a modestly high response rate of 40%.

The study will initially enroll 10 evaluable patients in each arm. If 0 or 1 of the 10 patients has a clinical response, then no further patients will be accrued. If 2 or more the first 10 patients have a response, then accrual continues to a total of 22 patients in each arm.

ELIGIBILITY:
* INCLUSION CRITERIA:

Status Update: Patients enrolled after Amendment G (version dated 08/16/2013), will be evaluated and compared to the first 13 patients by the study statistician and the Principal Investigator.

* Patients must have histologically confirmed metastatic alveolar soft part sarcoma that is not curable by surgery. Diagnosis of malignancy must be confirmed by the department of pathology at the institution where the patient is enrolled prior to patient enrollment.
* Patients must show evidence of objective disease progression per Response Evaluation Criteria in Solid Tumors (RECIST)v 1 on scans within the 6-month period immediately preceding enrollment. Both scans used to determine disease progression should have been obtained within this 6-month period.
* Patients with newly diagnosed, unresectable, metastatic, and measurable alveolar soft part sarcoma (ASPS) who show clinical evidence of disease progression (including history and increasing physical symptoms) will also be eligible. On-study documentation will include a physician's rationale that supports evidence of clinical disease progression (i.e., increasing tumor pain).
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
* Any prior therapy must have been completed greater than or equal to 4 weeks prior to enrollment on protocol and the participant must have recovered to eligibility levels from prior toxicity. Patients should be at least 6 weeks out from nitrosoureas and mitomycin C. Prior radiation should have been completed greater than or equal to 4 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels. Patients who have had prior monoclonal antibody therapy must have completed that therapy at least 3 half-lives of the antibody or 6 weeks ago. Patients who have received more than a cumulative dose of 350 mg/m(2) of doxorubicin may be enrolled at the discretion of the Coordinating Center PI after consultation with a cardiologist and if screening echocardiogram is normal.
* Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study (also referred to as an early Phase I study or pre-Phase I study where a sub-therapeutic dose of drug is administered) at the Coordinating Center principal investigator (PI's) discretion and should have recovered to eligibility levels from any toxicities.
* Patients with no prior therapy are eligible, provided they have metastatic disease that is not curable by surgery.
* Age greater than or equal to 16 years. Patients age 16-17 years are eligible only if they have a BSA greater than or equal to 1.7 m(2) or weigh greater than or equal to 60 kg.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin greater than or equal to 9 g/dL
  * total serum bilirubin within normal institutional limits
  * aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT) less than or equal to 2.5 times institutional upper limit of normal
  * creatinine within normal institutional limits

OR

* creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels above institutional normal
* QT corrected for heart rate (QTc) <480 msec (with Bazett's correction) in screening electrocardiogram.
* The following groups of patients are eligible after consultation with a cardiologist and at the Coordinating Center PI's discretion, provided they have New York Heart Association Class II (NYHA) cardiac function on baseline echocardiogram (ECHO):
* those with a history of Class II heart failure who are asymptomatic on treatment
* those with prior anthracycline exposure greater than a cumulative dose of 350 mg/m(2)
* those who have received central thoracic radiation that included the heart in the radiotherapy port.
* Patients must have blood pressure (BP) no greater than 140 millimeters of mercury (mmHg) (systolic) and 90 mmHg (diastolic) for eligibility. Initiation or adjustment of BP medication is permitted prior to study entry provided that the BP reading prior to enrollment is no greater than 140/90 mmHg.
* Left ventricular ejection fraction (LVEF) greater than or equal to institutional lower limit of normal.
* Because sunitinib is metabolized primarily by the cytochrome P450 3A4 (CYP3A4) liver enzyme, strong CYP3A4 inhibitors are not permitted within 7 days before and during the study, and strong CYP3A4 inducers are not permitted within 12 days before and during the study. A list of drugs that may interact with the cytochrome P450 system is included in Appendix C. Every effort should be made to switch patients taking such agents or substances to other medications 1 week prior to starting therapy, particularly patients with brain metastases who are taking enzyme- inducing anticonvulsant agents (Appendix D). Patients who require potent CYP3A4 inducers or inhibitors and cannot switch medications must have their case reviewed by the Coordinating Center PI and may be enrolled only after discussion with and agreement from the Coordinating Center PI. Current clinical studies with cediranib have not found clinically significant effects on cediranib pharmacokinetic (PK) with co-administration of CYP3A4 inducers or inhibitors. Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics (PK) of cediranib will be determined following review of their case by the Coordinating Center PI.
* Both study agents have been shown to terminate fetal development in the rat, as expected for a process dependent on VEGF signaling. For this reason, women of childbearing potential must have a negative pregnancy test prior to study entry.

Women of child-bearing potential and men must agree to use two reliable forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 2 months following study drug discontinuation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

* Patients who are nursing infants: because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated with the study agents.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must be able to swallow whole tablets and capsules.

EXCLUSION CRITERIA:

* Patients must not have received prior treatment with any VEGF receptor tyrosine kinase inhibitor (e.g., cediranib, sunitinib, pazopanib, sorafenib); however, prior treatment with bevacizumab is allowed.
* Patients may not be receiving any other investigational agents.
* Major surgery within 4 weeks prior to entry into the study, or a surgical incision that is not fully healed.
* History of familial long QT syndrome, or use of medications that may cause QTc interval prolongation.
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible.
* Warfarin and its derivatives are not allowed. Patient can be receiving low molecular weight heparin if clinically indicated.
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow, retain, and/or absorb the drug are excluded.
* Patients with any of the following conditions are excluded: serious or non-healing wound, ulcer; history of abdominal fistula, gastrointestinal perforation, or intra - abdominal abscess within 28 days of treatment; coronary/peripheral artery bypass graft or stenting within the past 12 months; or cerebrovascular accident (CVA) or transient ischemic attack within the past 12 months.
* Greater than 2+ proteinuria on two consecutive dipsticks taken no less than 1 week apart or 24-hour urine protein of > 1 g. Patients with < 2+ proteinuria are eligible following initial determination by urinalysis within 1 week prior to enrollment and do not need the urinalysis repeated.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for PK interactions with cediranib or sunitinib. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-07-18 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2026-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Requests for all collected individual participant data (IPD) data from clinical trials, conducted under a binding collaborative agreement between national Cancer Institute (NCI)/Division of Cancer Treatment and Diagnosis (DCTD) and a pharmaceutical/biotechnology company, that are not under Data and Safety Monitoring Board (DSMB) monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI Experimental Therapeutics Clinical Trials Network (ETCTN) Director in conjunction with the NCI/DCTD Regulatory Affairs Branch).

REFERENCES:
- [Background] Anderson ME, Hornicek FJ, Gebhardt MC, Raskin KA, Mankin HJ. Alveolar soft part sarcoma: a rare and enigmatic entity. Clin Orthop Relat Res. 2005 Sep;438:144-8. doi: 10.1097/01.blo.0000180049.50832.4a. PMID 16131883
- [Background] Azizi AA, Haberler C, Czech T, Gupper A, Prayer D, Breitschopf H, Acker T, Slavc I. Vascular-endothelial-growth-factor (VEGF) expression and possible response to angiogenesis inhibitor bevacizumab in metastatic alveolar soft part sarcoma. Lancet Oncol. 2006 Jun;7(6):521-3. doi: 10.1016/S1470-2045(06)70729-X. No abstract available. PMID 16750504
- [Background] Bello CL, Sherman L, Zhou J, Verkh L, Smeraglia J, Mount J, Klamerus KJ. Effect of food on the pharmacokinetics of sunitinib malate (SU11248), a multi-targeted receptor tyrosine kinase inhibitor: results from a phase I study in healthy subjects. Anticancer Drugs. 2006 Mar;17(3):353-8. doi: 10.1097/00001813-200603000-00015. PMID 16520665
- [Result] Nguyen J, Takebe N, Kummar S, Razak A, Chawla SP, George S, Patel SR, Keohan ML, Movva S, O'Sullivan Coyne G, Do K, Juwara L, Augustine B, Steinberg SM, Kuhlmann L, Ivy SP, Doroshow JH, Chen AP. Randomized Phase II Trial of Sunitinib or Cediranib in Alveolar Soft Part Sarcoma. Clin Cancer Res. 2023 Apr 3;29(7):1200-1208. doi: 10.1158/1078-0432.CCR-22-2145. PMID 36302173
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0200.html

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD2171 (Cediranib) 30 mg: Treatment assignment code 1. Part I: Participants will be randomized to receive cediranib (30 mg) orally, once a day, in 28-day cycles. Part I is a two-stage design in which 10 participants are initially enrolled in each arm. If 0 or 1 of the 10 participants has a clinical response, then no further participants will be accrued. That treatment arm will be closed to the accrual of new participants and the crossover of participants who progressed on the other agent. If 2 or more the first 10 participants have a response, then accrual would continue until a total of 22 participants have enrolled in that arm. Part II: At the time of disease progression (documented by Response Evaluation Criteria in Solid Tumors (RECIST v1), participants will cross over to the other treatment arm after a 2-week wash-out period (unless the other arm has been closed due to inadequate activity or unacceptable toxicity).
- AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg: Treatment assignment code 1 followed by treatment assignment code 2. Part I: Participants will be randomized to receive cediranib (30 mg) or sunitinib malate (37.5 mg) orally, once a day, in 28-day cycles. Part I is a two-stage design in which 10 participants are initially enrolled in each arm. If 0 or 1 of the 10 participants has a clinical response, then no further participants will be accrued. That treatment arm will be closed to the accrual of new participants and the crossover of participants who progressed on the other agent. If 2 or more the first 10 patients have a response, then accrual would continue until a total of 22 participants have enrolled in that arm. Part II: At the time of disease progression (documented by Response Evaluation Criteria in Solid Tumors (RECIST v1), participants will cross over to the other treatment arm after a 2-week wash-out period (unless the other arm has been closed due to inadequate activity or unacceptable toxicity).
- Sunitinib Malate 37.5 mg: Treatment assignment code 2. Part I: Participants will be randomized to receive sunitinib malate (37.5 mg) orally, once a day, in 28-day cycles. Part I is a two-stage design in which 10 participants are initially enrolled in each arm. If 0 or 1 of the 10 participants has a clinical response, then no further participants will be accrued. That treatment arm will be closed to the accrual of new participants and the crossover of participants who progressed on the other agent. If 2 or more the first 10 participants have a response, then accrual would continue until a total of 22 participants have enrolled in that arm. Part II: At the time of disease progression (documented by Response Evaluation Criteria in Solid Tumors (RECIST v1), patients will cross over to the other treatment arm after a 2-week wash-out period (unless the other arm has been closed due to inadequate activity or unacceptable toxicity).
- Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg: Treatment assignment code 2 followed by treatment assignment code 1. Part I: Participants will be randomized to receive cediranib (30 mg) or sunitinib malate (37.5 mg) orally, once a day, in 28-day cycles. Part I is a two-stage design in which 10 patients are initially enrolled in each arm. If 0 or 1 of the 10 participants has a clinical response, then no further participants will be accrued. That treatment arm will be closed to the accrual of new participants and the crossover of participants who progressed on the other agent. If 2 or more the first 10 participants have a response, then accrual would continue until a total of 22 participants have enrolled in that arm. Part II: At the time of disease progression (documented by Response Evaluation Criteria in Solid Tumors (RECIST v1), participants will cross over to the other treatment arm after a 2-week wash-out period (unless the other arm has been closed due to inadequate activity or unacceptable toxicity).
Period: Part I
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Started | 7 | 9 | 5 | 13
Restaging | 6 | 9 | 4 | 12
Pharmacokinetic sampling | 2 | 6 | 0 | 0
Completed | 7 | 9 | 5 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Washout - 2 Weeks
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Started | 0 | 9 | 0 | 13
Completed | 0 | 9 | 0 | 13
Not Completed | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Started | 0 | 9 | 0 | 13
Restaging | 0 | 9 | 0 | 13
Pharmacokinetic sampling | 0 | 0 | 0 | 7
Completed | 0 | 9 | 0 | 13
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg | Total
Number analyzed (Participants) | 7 | 9 | 5 | 13 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1 | 2
  Between 18 and 65 years | 7 | 8 | 5 | 11 | 31
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.67 (11.03) | 26.6 (6.03) | 30.88 (17.74) | 32.87 (13.72) | 29.64 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 7
  Male | 5 | 7 | 4 | 11 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 5 | 9 | 4 | 13 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 1 | 5 | 0 | 4 | 10
  White | 6 | 1 | 4 | 5 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 5 | 13 | 34

OUTCOME MEASURES:

1. Primary Outcome: Part I: Objective Response Rate (ORR) of Single-agent Cediranib in Participants With Advanced Alveolar Soft Part Sarcoma (ASPS)
Description: Objective response rate is the combined partial and complete response rate, with those terms defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response is disappearance of all non-target lesion and normalization of tumor marker level. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of the LD.
Time Frame: Time on treatment (an average of 497 days or 16 months)
Population: A total of 15/34 participants were analyzed: 15/16 participants who received cediranib in Part I were analyzed (1 participant was not evaluable for response).
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg
Number analyzed (Participants) | 6 | 9
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 1

2. Primary Outcome: Part I: Objective Response Rate (ORR) of Single-agent Sunitinib in Participants With Advanced Alveolar Soft Part Sarcoma (ASPS)
Description: as for outcome 1
Time Frame: Time on treatment (an average of 497 days or 16 months)
Population: A total of 14/34 participants were analyzed: 14/18 participants who received sunitinib in Part I were analyzed (4 participants who received sunitinib were not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 4 | 10
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 1

3. Primary Outcome: Part II: Objective Response Rate (ORR) of Sunitinib in Participants Who Progress on the Cediranib Arm During Part I
Description: as for outcome 1
Time Frame: Time on treatment (an average of 497 days or 16 months)
Population: A total of 9/34 participants were analyzed: 9/9 participants who received sunitinib in Part II were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 0

4. Primary Outcome: Part II: Objective Response Rate (ORR) of Cediranib in Participants Who Progress on the Sunitinib Arm During Part I
Description: as for outcome 1
Time Frame: Time on treatment (an average of 497 days or 16 months)
Population: A total of 10/34 participants were analyzed: 10/13 participants who received cediranib in Part II were analyzed (3 participants were not evaluable for response).
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 10
Participants
  Complete Response | 0
  Partial Response | 1

5. Secondary Outcome: Maximum Observed Plasma Concentration of Cediranib
Description: Pharmacokinetic analysis was performed on blood samples from participants on cediranib (both upfront therapy and following cross-over). Human plasma samples were analyzed using a validated liquid chromatography-mass spectrometry (LC-MS) method and the maximum observed analyte concentration in plasma will be reported. No sampling or analysis will be done for participants receiving sunitinib.
Time Frame: Before first dose on Cycle 1 day 15, Cycle 2 Day 1, Cycle 3 Day 1, and Cycle 4 Day 1 (each cycle is 28 days)
Population: A total of 15/34 participants were analyzed: 15/29 participants who received cediranib in either Part I or Part II were analyzed.
Measure: Mean (Full Range); unit: Nanomolar
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 2 | 6 | 7
Nanomolar | 108 [47 to 168] | 115 [36 to 219] | 126 [54 to 194]

6. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS) at 24 Weeks for Participants Receiving Single-agent Cediranib and Single-agent Sunitinib Malate in Participants With Advanced ASPS During Part I
Description: 24-week PFS is defined as the probability of participants remaining alive and progression-free at 24 weeks after the start of treatment. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 24 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 7 | 9 | 5 | 13
Percentage of participants | 62.5 [29.5 to 76.2] | 62.5 [29.5 to 76.2] | 50.0 [25.9 to 70.1] | 50.0 [25.9 to 70.1]

7. Secondary Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, an average of 523 days
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 7 | 9 | 5 | 13
Participants | 7 | 9 | 4 | 13

8. Other Pre Specified Outcome: Best Overall Response During Part I for Participants Who Were Not Newly Diagnosed
Description: Best overall response is the best response recorded from the start of the treatment until disease progression/recurrence. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response is disappearance of all non-target lesion and normalization of tumor marker level. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of the LD. Progression is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Stable disease is neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: Time on treatment (an average of 497 days or 16 months)
Population: A total of 11/34 participants were analyzed: of the 14 participants who were not newly diagnosed, 2 participants randomized to receive sunitinib and 1 participant randomized to receive cediranib in Part I were not evaluable for response, leaving only 11 reportable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 0 | 3 | 1 | 7
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 1
  Stable Disease | 0 | 3 | 1 | 5
  Progressive Disease | 0 | 0 | 0 | 1

9. Other Pre Specified Outcome: Percentage of Participants With Progression-free Survival (PFS) at 24 Weeks During Part I for Participants Who Were Not Newly Diagnosed
Description: 24-week PFS is defined as the probability of patients remaining alive and progression-free at 24 weeks after the start of treatment. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: 24 weeks
Population: A total of 14/34 participants were analyzed. 20 participants not analyzed were newly diagnosed. The outcome is for non-newly diagnosed participants only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 1 | 3 | 2 | 8
Percentage of participants | 50.0 [5.8 to 84.5] | 50.0 [5.8 to 84.5] | 40.0 [12.3 to 67.0] | 40.0 [12.3 to 67.0]

10. Other Pre Specified Outcome: Best Overall Response During Part II for Participants Who Were Not Newly Diagnosed
Description: as for outcome 8
Time Frame: Time on treatment (an average of 497 days or 16 months)
Population: A total of 10/34 participants were analyzed: of the 11 participants who were not newly diagnosed and participated in Part II of the trial, 1 participant (who was randomized to receive sunitinib in Part I and then crossed over to receive cediranib in Part II) was not evaluable for response, leaving only 10 reportable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 0 | 3 | 0 | 7
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 1
  Stable Disease | 0 | 2 | 0 | 3
  Progressive Disease | 0 | 1 | 0 | 2
  Not Scanned | 0 | 0 | 0 | 1

11. Other Pre Specified Outcome: Percentage of Participants With Progression-free Survival (PFS) at 24 Weeks During Part II for Participants Who Were Not Newly Diagnosed
Description: as for outcome 9
Time Frame: 24 weeks
Population: 11/34 participants were analyzed: all 11 participants who were not newly diagnosed and participated in Part II of the trial were analyzed. 20 participants were not analyzed as they were newly diagnosed and this outcome is for non-newly diagnosed participants only. In addition, 3 participants who were not newly diagnosed did not participate in Part II of the trial, leaving 11 participants who were not newly diagnosed and who participated in Part II of the trial, for whom this outcome is reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZD2171 (Cediranib) 30 mg | AZD2171 (Cediranib) 30 mg Followed by Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg | Sunitinib Malate 37.5 mg Followed by AZD2171 (Cediranib) 30 mg
Number analyzed (Participants) | 0 | 3 | 0 | 8
percentage of participants |  | 33.3 [0.9 to 77.4] |  | 57.1 [17.2 to 83.7]

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, an average of 523 days
Description: 23 subjects in the Cediranib Group were first treated with Cediranib before crossing over to receive Sunitinib; and 6 subjects received Cediranib treatment only.
  23 subjects in the Sunitinib Group were first treated with Cediranib before receiving Sunitinib; and 4 subjects received Sunitinib treatment only.
  The "Number of Subjects Affected/Number of Events" for serious and other adverse events is derived from specific courses of treatment where each agent was administered for each subject.
Groups:
- Sunitinib Malate 37.5 mg: Treatment assignment code 2. Part I: Participants will be randomized to receive sunitinib malate (37.5 mg) orally, once a day, in 28-day cycles. Part I is a two-stage design in which 10 participants are initially enrolled in each arm. If 0 or 1 of the 10 participants has a clinical response, then no further participants will be accrued. That treatment arm will be closed to the accrual of new participants and the crossover of participants who progressed on the other agent. If 2 or more the first 10 participants have a response, then accrual would continue until a total of 22 participants have enrolled in that arm. Part II: At the time of disease progression (documented by Response Evaluation Criteria in Solid Tumors (RECIST v1), patients will cross over to the other treatment arm after a 2-week wash-out period (unless the other arm has been closed due to inadequate activity or unacceptable
Arm/Group | AZD2171 (Cediranib) 30 mg | Sunitinib Malate 37.5 mg
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/27
Serious Adverse Events (participants affected / at risk) | 7/29 | 7/27
Other Adverse Events (participants affected / at risk) | 28/29 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD2171 (Cediranib) 30 mg (N=29) | Sunitinib Malate 37.5 mg (N=27)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, perianal abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, Candidal Infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, Domestic assault (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, brain metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pregnancy, puerperium and perinatal conditions - Other, Pregnancy of spouse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD2171 (Cediranib) 30 mg (N=29) | Sunitinib Malate 37.5 mg (N=27)
Abdominal pain (Gastrointestinal disorders) | 13 (20) | 3 (3)
Alanine aminotransferase increased (Investigations) | 12 (20) | 11 (22)
Alkaline phosphatase increased (Investigations) | 7 (8) | 4 (6)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 10 (26) | 15 (35)
Anorexia (Metabolism and nutrition disorders) | 13 (13) | 7 (7)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 16 (31) | 14 (25)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 5 (17) | 4 (4)
Blurred vision (Eye disorders) | 0 (0) | 4 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
CPK increased (Investigations) | 1 (2) | 2 (3)
Cheilitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (10) | 9 (10)
Corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Creatinine increased (Investigations) | 6 (14) | 5 (9)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 22 (54) | 17 (30)
Dizziness (Nervous system disorders) | 8 (12) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 6 (6)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (4)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 4 (4)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (2) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Eye disorders - Other, Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, bright spots/halo (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fatigue (General disorders) | 10 (14) | 11 (19)
Fever (General disorders) | 4 (4) | 3 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3)
Flu like symptoms (General disorders) | 1 (4) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrointestinal disorders - Other, Anal Abscess (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Gastrointestinal disorders - Other, abdominal cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Oral sensitivity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, perianal abscess (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, left shoulder pain (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, non cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 8 (17)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 2 (3)
Hemoglobinuria (Renal and urinary disorders) | 2 (3) | 4 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 8 (10) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (10) | 4 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 18 (280) | 16 (149)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (12) | 5 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (9) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 9 (15) | 4 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5) | 5 (14)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Hypothyroidism (Endocrine disorders) | 8 (9) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Infections and infestations - Other, dacryocystitis (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, right inner thigh cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Other, yeast infection (Infections and infestations) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, Broken nose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, Gait change due to fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, Right pathological fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Investigations - Other, Decreased White Blood Cell Count (Investigations) | 1 (1) | 0 (0)
Investigations - Other, Increased AST-SGOT (Investigations) | 1 (1) | 0 (0)
Investigations - Other, Increased BUN (Investigations) | 1 (1) | 0 (0)
Investigations - Other, Increased Phosphorus (Investigations) | 1 (1) | 0 (0)
Investigations - Other, Increased TSH (Investigations) | 1 (1) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 13 (28) | 12 (38)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (5) | 11 (15)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Left hip pain from fall intermittent (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) — Musculoskeletal and connective tissue disorder - Other, rib and bilateral knee pain
Musculoskeletal and connective tissue disorder - Other, Right hip and thigh pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (15) | 10 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nervous system disorders - Other, Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (14) | 18 (86)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (6) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9) | 4 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (10) | 10 (18)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 3 (3) | 2 (3)
Periorbital edema (Eye disorders) | 0 (0) | 2 (2)
Pharyngeal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 8 (18) | 14 (33)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pregnancy, puerperium and perinatal conditions - Other, Pregnancy of spouse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 9 (28) | 10 (22)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5) | 5 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Reproductive system and breast disorders - Other, Painful prolonged erection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, scrotal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, patient noted a "runny nose" (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 7 (13) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (3)
Skin and subcutaneous tissue disorders - Other, Bl feet corns (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Hair pigment change (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Skin and subcutaneous tissue disorders - Other, specify Mouth ulcers
Skin and subcutaneous tissue disorders - Other, Small scabs to buttocks (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, change in hair color (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, eschar on left gluteal area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, finger tip color change (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, graying hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, hair hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (11)
Skin infection (Infections and infestations) | 3 (4) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Thyroid stimulating hormone increased (Endocrine disorders) | 1 (2) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 4 (4)
Upper respiratory infection (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (16) | 4 (6)
Weight gain (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 9 (15) | 2 (2)
White blood cell decreased (Investigations) | 8 (17) | 20 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT01391962/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT01391962/ICF_001.pdf